CLINICAL TRIAL: NCT03469531
Title: Efficacy and Safety of Nimotuzumab Combined With Radiotherapy and Concurrently Cisplatin in Patients With Stage IIB-IVA Cervical Squamous Cell Carcinoma
Brief Title: Study of Nimotuzumab Combined With Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-ZLZX-002
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-02

CONDITIONS: Neoplasms; Cervical Adenosquamous Cell Carcinoma; Cervical Squamous Cell Carcinoma in Situ; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
Keywords: Cervical Cancer; Radiation Therapy; Chemotherapy; Nimotuzumab; Cisplatin
MeSH Terms: conditions — Neoplasms; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — nimotuzumab; Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients receive nimotuzumab combined with cisplatin and undergo external-beam radiation and brachytherapy as the patients in experimental group.
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Radiation: external-beam radiation; Radiation: brachytherapy
- control group (Active Comparator): Patients receive cisplatin and undergo external-beam radiation and brachytherapy as the patients in control group.
  Interventions: Drug: Cisplatin; Radiation: external-beam radiation; Radiation: brachytherapy

INTERVENTIONS:
Drug: Nimotuzumab — Patients receive nimotuzumab IV over 90 minutes on days 1, 8, 15, 22, 29, 36,43.
  Other Names: EGFR monoclonal antibody
  Arms: experimental group
Drug: Cisplatin — Patients undergo cisplatin, 25-40 mg/m2 a week for 4 or 5weeks
  Other Names: Cisplatin injection
Radiation: external-beam radiation — Patients undergo pelvic EBRT once daily, 5 days a week, for 5 weeks for a total of 45-50.4Gy
  Other Names: pelvic EBRT
Radiation: brachytherapy — high-dose rate brachytherapy,6Gy once weekly,for a total of 24-30Gy
  Other Names: high-dose rate brachytherapy

SUMMARY:
The purpose of this phase II trial is to determine the feasibility and efficacy of nimotuzumab combined with concurrent chemoradiotherapy for initially inoperable locally advanced cervical squamous cell carcinoma.

DETAILED DESCRIPTION:
This phase II trial is studying how well giving nimotuzumab together with radiation therapy and cisplatin works in treating patients with previously untreated locally advanced cervical cancer. Monoclonal antibodies, such as nimotuzumab, a humanized anti-epidermal growth factor receptor (EGFR) monoclonal antibody that is approved in many countries for the treatment of EGFR-positive cancers. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Nimotuzumab also stop the growth of cervical cancer by increasing the effect of chemotherapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving nimotuzumab together with radiation therapy and cisplatin may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers will sign the informed consent.
* Histologically confirmed squamous cell of the uterine cervix, EGFR(+).
* The FIGO stage (IIB-IVA) and was not available for surgical treatment.
* There is at least one tumor lesion that is measurable by RECIST.
* During the study, contraception should be ensured.
* Karnofsky performance status >60.
* WBC >= 3,000/mm^3
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* INR < 1.5
* Total bilirubin =< 1.5 mg/dL
* Serum creatinine =< 1.5 mg/dL
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Serum calcium =< 1.3 times ULN
* Hemoglobin >= 9g/dL (transfusion allowed)

Exclusion Criteria:

* Positive para-aortic lymph nodes or positive lymph nodes beyond pelvic
* Prior invasive malignancy (except nonmelanomatous skin cancer)
* Contraindication of chemotherapy;
* Rare pathological subtype;
* Cervical cancer patients underwent hysterectomy, laparoscopic surgery or systemic chemotherapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
progress free survival rate | 3 years
  The rate of patient without progress disease in 3 years after treatment

SECONDARY OUTCOMES:
Overall survival rate | 3 years
  The rate of patient alive in 3 years after treatment
Local area control rate. | 3 years
  The rate of patient without recurrence in 3 years after treatment
No distant metastatic survival. | 3 years
  The rate of patient without metastatic disease in 3 years after treatment
objective response rate | 3 years
  the percentage of patients who experienced complete or partial cancer shrinkage or disappearance after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: junguo bu, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No